CLINICAL TRIAL: NCT00922896
Title: A Phase II Trial of Erlotinib in Combination With Gemcitabine and Cisplatin in Metastatic Pancreatic Cancer
Brief Title: Trial of Erlotinib, Gemcitabine and Cisplatin in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: Dong-A University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Jung Hun Kang, Associate Professor, Gyeongsang National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gyeongsang-001
Record Dates: First submitted 2009-06-02; First posted 2009-06-17 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Gemcitabine; Cisplatin; Erlotinib
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Cisplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GPE (Experimental): Gemcitabine-Cisplatin-Erlotinib
  Interventions: Drug: Gemcitabine, Cisplatin, Erlotinib (Tarceva)

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin, Erlotinib (Tarceva) — * Erlotinib 100 mg po q d daily AND
  * Gemcitabine 1000 mg/m² with 250 mL of normal saline intravenously infusion over 30 mins on Day 1, 8
  * Cisplatin 25 mg/m2 with 150 mL of normal saline intravenously infusion over 60 mins on D1,8
  Every 3 weeks

SUMMARY:
The purpose of this study is to determine the response rate of gemcitabine, cisplatin and erlotinib in metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18
* Younger than 75
* ECOG performance status 0 or 1
* Histologically confirmed adenocarcinoma of the pancreas
* Metastatic pancreatic cancer
* No prior chemotherapy for metastatic pancreatic cancer
* A patient with at least one measurable primary lesion of which the diameter is confirmed to be 10mm in Spiral CT or multidetector CT (MD CT)

Exclusion Criteria:

* A patient with no measurable disease
* A patient who received previous palliative chemotherapy for pancreatic cancer
* A patient with locally advanced pancreatic cancer
* A patient who received adjuvant chemotherapy for pancreatic cancer within 1 year
* A patient with previous active or passive immunotherapy
* A pregnant or lactating patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess the response rate associated with gemcitabine, erlotinib and cisplatin in patients with advanced pancreatic cancer | Clinically assessed every cycle (month) and radiologically assessed every 2 cycles (6 weeks) with CT scan

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Dong-A University Hospital, Busan
  - Gyeongsang Unversity Hospital, Jinju
  - Chung-Ang University Hospital, Seoul

REFERENCES:
- [Derived] Hwang IG, Jang JS, Oh SY, Lee S, Kwon HC, Lee GW, Go S, Kang MH, Cha YJ, Kang JH. A phase II trial of Erlotinib in combination with gemcitabine and cisplatin in advanced pancreatic cancer. Invest New Drugs. 2012 Dec;30(6):2371-6. doi: 10.1007/s10637-012-9792-z. PMID 22302349